CLINICAL TRIAL: NCT02501629
Title: A Phase 3, 24-Week Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy and Safety Study of Reslizumab Subcutaneous Dosing (110 mg Every 4 Weeks) in Patients With Oral Corticosteroid Dependent Asthma and Elevated Blood Eosinophils
Brief Title: An Efficacy and Safety Study of Reslizumab Subcutaneous in Patients With Oral Corticosteroid Dependent Asthma and Elevated Blood Eosinophils
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C38072-AS-30027; 2015-001580-39 (EudraCT Number)
Record Dates: First submitted 2015-07-14; First posted 2015-07-17 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma; Elevated Blood Eosinophils; Oral Corticosteroid Dependence
Keywords: Asthma; Elevated Blood Eosinophils; Oral corticosteroid dependence; Reslizumab
MeSH Terms: conditions — Asthma | interventions — reslizumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reslizumab 110 mg (Experimental): Reslizumab was administered by subcutaneous injection (sc) in a dosage of 110 mg (1.0 mL) every 4 weeks for a total of six doses.
  Interventions: Drug: Reslizumab; Drug: Non-Oral Corticosteroid (non-OCS) Asthma Medication; Drug: Oral Corticosteroid (OCS)
- Placebo (Placebo Comparator): Matching placebo was administered by subcutaneous injection (sc) 1.0 mL every 4 weeks for a total of six doses.
  Interventions: Drug: Placebo; Drug: Non-Oral Corticosteroid (non-OCS) Asthma Medication; Drug: Oral Corticosteroid (OCS)

INTERVENTIONS:
Drug: Reslizumab — Reslizumab 110 mg was administered by qualified study personnel as subcutaneous injections in the upper arm(s) once every 4 weeks for a total of 6 doses. Drug was supplied in pre-filled syringes.
  Other Names: CEP38072
  Arms: Reslizumab 110 mg
Drug: Placebo — Placebo was administered by qualified study personnel as subcutaneous injections in the upper arm(s) once every 4 weeks for a total of 6 doses. Drug was supplied in pre-filled syringes.
  Arms: Placebo
Drug: Non-Oral Corticosteroid (non-OCS) Asthma Medication — Participants continue using their non-OCS background asthma medications without change during the study's treatment period.
Drug: Oral Corticosteroid (OCS) — After screening and prior to study start, the participant's OCS dose was adjusted to determine the minimal effective OCS requirement.

SUMMARY:
The primary objective of the study is to determine the ability of reslizumab administered by subcutaneous injection to produce a corticosteroid-sparing effect in patients with oral corticosteroid (OCS)-dependent asthma and elevated blood eosinophils, without loss of asthma control.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is male or female, 12 years of age and older, with a previous diagnosis of asthma.
2. Written informed consent is obtained.
3. The patient requires daily maintenance dose of prednisone or equivalent for asthma of between 5 and 40 mg during the 3 months prior to screening.
4. The patient has a documented elevated blood eosinophils at screening or during the previous 12 months.
5. The patient has required high dose ICS plus another asthma controller for at least 6 months prior to screening.
6. The patient has FEV1 reversibility to inhaled SABA or historical reversibility within the previous 24 months.

   * Other criteria may apply, please contact the investigator for more information.

Exclusion Criteria:

1. The patient has any clinically significant, uncontrolled medical condition that would interfere with the study schedule or procedures and interpretation of efficacy results or would compromise the patient's safety.
2. The patient has another confounding underlying lung disorder.
3. The patient has a known hypereosinophilic syndrome.
4. The patient has a history of any malignancy within 5 years of the screening visit, except for treated and cured non-melanoma skin cancers.
5. The patient is pregnant or intends to become pregnant during the study or is lactating.
6. The patient required treatment for an asthma exacerbation within 4 weeks of screening.
7. The patient is a current smoker or has a smoking history ≥10 pack-years.
8. The patient is currently using any systemic immunosuppressive or immunomodulatory biologic except maintenance OCS for the treatment of asthma.
9. The patient participated in a clinical study within 30 days or 5 half-lives of the investigational drug before screening, whichever is longer.
10. The patient was previously exposed to benralizumab within 12 months of screening.
11. The patient was previously exposed to reslizumab.
12. The patient has a history of immunodeficiency disorder including human immunodeficiency virus.
13. The patient has current suspected drug and/or alcohol abuse.
14. The patient has had an active helminthic parasitic infection or was treated for one within 6 months of screening.
15. The patient has a history of allergic reactions or hypersensitivity to any component of the study drug.

    * Other criteria may apply, please contact the investigator for more information.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (127):
- United States (26):
  - Teva Investigational Site 13357, Bakersfield, California
  - Teva Investigational Site 13365, Long Beach, California
  - Teva Investigational Site 13371, Clermont, Florida
  - Teva Investigational Site 13351, Homestead, Florida
  - Teva Investigational Site 13342, Kissimmee, Florida
  - Teva Investigational Site 13344, Miami, Florida
  - Teva Investigational Site 13372, Miami, Florida
  - Teva Investigational Site 13354, Pembroke Pines, Florida
  - Teva Investigational Site 13343, Saint Cloud, Florida
  - Teva Investigational Site 13368, Sebring, Florida
  - Teva Investigational Site 13346, Tampa, Florida
  - Teva Investigational Site 13367, Chicago, Illinois
  - Teva Investigational Site 13363, Normal, Illinois
  - Teva Investigational Site 13345, Michigan City, Indiana
  - Teva Investigational Site 13348, Lenexa, Kansas
  - Teva Investigational Site 13362, Biloxi, Mississippi
  - Teva Investigational Site 13350, St Louis, Missouri
  - Teva Investigational Site 13352, St Louis, Missouri
  - Teva Investigational Site 13356, New York, New York
  - Teva Investigational Site 13349, Cincinnati, Ohio
  - Teva Investigational Site 13370, Edmond, Oklahoma
  - Teva Investigational Site 13347, Oklahoma City, Oklahoma
  - Teva Investigational Site 13366, Charleston, South Carolina
  - Teva Investigational Site 13377, Dallas, Texas
  - Teva Investigational Site 13369, Houston, Texas
  - Teva Investigational Site 13358, Fairfax, Virginia
- Argentina (10):
  - Teva Investigational Site 20059, Buenos Aires
  - Teva Investigational Site 20058, Buenos Aires
  - Teva Investigational Site 20056, Buenos Aires
  - Teva Investigational Site 20057, Buenos Aires
  - Teva Investigational Site 20052, Córdoba
  - Teva Investigational Site 20055, Mendoza
  - Teva Investigational Site 20050, Mendoza
  - Teva Investigational Site 20087, Rosario
  - Teva Investigational Site 20051, San Miguel de Tucumán
  - Teva Investigational Site 20066, San Rafael
- Australia (6):
  - Teva Investigational Site 78089, Bedford Park
  - Teva Investigational Site 78092, Box Hill
  - Teva Investigational Site 78097, Frankston
  - Teva Investigational Site 78093, Kent Town
  - Teva Investigational Site 78090, Nedlands
  - Teva Investigational Site 78091, New Lambton
- Belgium (2):
  - Teva Investigational Site 37059, Brussels
  - Teva Investigational Site 37058, Gembloux
- Czechia (2):
  - Teva Investigational Site 54133, Břeclav
  - Teva Investigational Site 54132, Jindřichův Hradec
- France (4):
  - Teva Investigational Site 35186, Le Kremlin-Bicêtre
  - Teva Investigational Site 35185, Lille
  - Teva Investigational Site 35189, Lyon
  - Teva Investigational Site 35187, Strasbourg
- Germany (8):
  - Teva Investigational Site 32621, Bad Wörishofen
  - Teva Investigational Site 32576, Berlin
  - Teva Investigational Site 32573, Berlin
  - Teva Investigational Site 32578, Berlin
  - Teva Investigational Site 32622, Frankfurt
  - Teva Investigational Site 32579, Hanover
  - Teva Investigational Site 32574, Leipzig
  - Teva Investigational Site 32580, Rostock
- Hungary (4):
  - Teva Investigational Site 51254, Csorna
  - Teva Investigational Site 51232, Dombóvár
  - Teva Investigational Site 51233, Hatvan
  - Teva Investigational Site 51253, Szombathely
- Israel (5):
  - Teva Investigational Site 80085, Haifa
  - Teva Investigational Site 80083, Jerusalem
  - Teva Investigational Site 80091, Kfar Saba
  - Teva Investigational Site 80084, Petah Tikva
  - Teva Investigational Site 80082, Rehovot
- Italy (2):
  - Teva Investigational Site 30152, Catanzaro
  - Teva Investigational Site 30154, Genova
- Mexico (11):
  - Teva Investigational Site 21106, Chihuahua City
  - Teva Investigational Site 21102, Distrito Federal
  - Teva Investigational Site 21104, Durango
  - Teva Investigational Site 21094, Guadalajara
  - Teva Investigational Site 21091, Guadalajara
  - Teva Investigational Site 21100, Guadalajara
  - Teva Investigational Site 21093, Guadalajara
  - Teva Investigational Site 21090, Mexico City
  - Teva Investigational Site 21103, Monterrey
  - Teva Investigational Site 21101, Monterrey
  - Teva Investigational Site 21105, Querétaro
- Netherlands (2):
  - Teva Investigational Site 38084, Leeuwarden
  - Teva Investigational Site 38085, Zwolle
- Poland (9):
  - Teva Investigational Site 53316, Gdansk
  - Teva Investigational Site 53318, Krakow
  - Teva Investigational Site 53319, Lodz
  - Teva Investigational Site 53321, Lodz
  - Teva Investigational Site 53322, Lubin
  - Teva Investigational Site 53320, Ostrów Wielkopolski
  - Teva Investigational Site 53358, Rzeszów
  - Teva Investigational Site 53317, Tarnów
  - Teva Investigational Site 53323, Wroclaw
- Russia (11):
  - Teva Investigational Site 50356, Barnaul
  - Teva Investigational Site 50417, Chelyabinsk
  - Teva Investigational Site 50385, Kemerovo
  - Teva Investigational Site 50382, Kemerovo
  - Teva Investigational Site 50384, Moscow
  - Teva Investigational Site 50383, Novosibirsk
  - Teva Investigational Site 50386, Novosibirsk
  - Teva Investigational Site 50357, Saint Petersburg
  - Teva Investigational Site 50418, Tomsk
  - Teva Investigational Site 50358, Tomsk
  - Teva Investigational Site 50419, Yekaterinburg
- South Korea (6):
  - Teva Investigational Site 87020, Goyang-si
  - Teva Investigational Site 87024, Jeonju
  - Teva Investigational Site 87025, Seongnam-si
  - Teva Investigational Site 87023, Seoul
  - Teva Investigational Site 87022, Seoul
  - Teva Investigational Site 87021, Seoul
- Spain (4):
  - Teva Investigational Site 31159, Barcelona
  - Teva Investigational Site 31161, Girona
  - Teva Investigational Site 31160, Valencia
  - Teva Investigational Site 31158, Valencia
- Ukraine (15):
  - Teva Investigational Site 58245, Dnipro
  - Teva Investigational Site 58238, Dnipropetrovsk
  - Teva Investigational Site 58240, Ivano-Frankivsk
  - Teva Investigational Site 58244, Kharkiv
  - Teva Investigational Site 58235, Kharkiv
  - Teva Investigational Site 58239, Kharkiv
  - Teva Investigational Site 58241, Kharkiv
  - Teva Investigational Site 58249, Kremenchuk
  - Teva Investigational Site 58248, Kyiv
  - Teva Investigational Site 58251, Kyiv
  - Teva Investigational Site 58237, Kyiv
  - Teva Investigational Site 58250, Kyiv
  - Teva Investigational Site 58243, Sumy
  - Teva Investigational Site 58246, Vinnytsia
  - Teva Investigational Site 58242, Zhaporizhzhya

REFERENCES:
- [Derived] Bernstein JA, Virchow JC, Murphy K, Maspero JF, Jacobs J, Adir Y, Humbert M, Castro M, Marsteller DA, McElhattan J, Hickey L, Garin M, Vanlandingham R, Brusselle G. Effect of fixed-dose subcutaneous reslizumab on asthma exacerbations in patients with severe uncontrolled asthma and corticosteroid sparing in patients with oral corticosteroid-dependent asthma: results from two phase 3, randomised, double-blind, placebo-controlled trials. Lancet Respir Med. 2020 May;8(5):461-474. doi: 10.1016/S2213-2600(19)30372-8. Epub 2020 Feb 14. PMID 32066536

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 273 patients with OCS-dependent severe eosinophilic asthma were screened, and 180 of these patients (at 78 centers) were considered eligible for enrollment. Three of the eligible patients were not randomized due to failure to meet randomization criteria.
Period: Overall Study
Arm/Group | Placebo | Reslizumab 110 mg
Started | 89 | 88
Completed (Participants who completed the 8-week follow-up visit or enrolled in NCT03052725) | 84 | 81
Not Completed | 5 | 7
Not completed — Death | 0 | 1
Not completed — Withdrawn from study by sponsor | 1 | 0
Not completed — Early termination by sponsor | 1 | 0
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Subject did not return to site | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent To Treat (ITT) Analysis Set: included all randomly assigned patients. Treatment grouping was based on the treatment to which patients were randomly assigned, regardless of which treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Reslizumab 110 mg | Total
Number analyzed (Participants) | 89 | 88 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (11.99) | 55.5 (12.72) | 54.3 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 60 | 117
  Male | 32 | 28 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 22 | 38
  Not Hispanic or Latino | 72 | 65 | 137
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 80 | 72 | 152
  Black or African American | 1 | 3 | 4
  Asian | 3 | 2 | 5
  American Indian or Alaska Native | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 4 | 8 | 12
Age Group [Count of Participants; unit: Participants]
  12 to <18 years | 1 | 0 | 1
  18 to <65 years | 74 | 63 | 137
  >=65 years | 14 | 25 | 39
Weight [Mean (Standard Deviation); unit: kg] | 82.69 (18.949) | 79.58 (21.390) | 81.14 (20.202)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.859 (6.3499) | 29.389 (8.0105) | 29.625 (7.2067)
Region Group [Count of Participants; unit: Participants]
  US/Canada | 10 | 9 | 19
  Europe | 58 | 47 | 105
  Other | 21 | 32 | 53
Oral Corticosteroid (OCS) Dose at Baseline [Mean (Standard Deviation); unit: mg] — The patient's previous OCS was standardized to an equivalent dose and regimen of prednisone to the nearest 2.5 mg daily. Prior to study, the dose was adjusted to identify the minimal effective OCS dose to control asthma symptoms without change to background asthma medications (non-OCS).
  mg | 10.37 (6.435) | 10.37 (6.807) | 10.37 (6.604)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction In Daily Oral Corticosteroid (OCS) Dose During Weeks 20-24 As Compared to the Optimized Dose At Baseline
Description: The primary endpoint was the 5-level categorized percent reduction in OCS dose during weeks 20 to 24 compared with the optimized dose at baseline. The primary analysis incorporated data from all randomized patients. Analysis of the primary and secondary variables related to categorical OCS dose reduction incorporated missing data as non-responders.
  No decrease indicates there was no decrease in OCS, loss of baseline asthma control during weeks 20 to 24, or discontinuation from study drug.
Time Frame: Baseline (Day 1), Weeks 20-24
Population: Intent to Treat (ITT) Analysis set; missing data are included as non-responders (no decrease).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 89 | 88
Participants
  90% to 100% | 20 | 18
  75% to <90% | 4 | 8
  50% to <75% | 8 | 13
  >0% to <50% | 9 | 7
  No decrease | 48 | 42
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 110 mg; The proportional odds ratio (reslizumab/placebo) was estimated from this model, representing the ratio of the odds of a patient outcome being in a higher OCS dose reduction category for reslizumab compared to placebo; Test type: Superiority; p = 0.468, proportional odds model — Significance at 0.05; factors for treatment group and randomization strata (age and OCS dose); baseline OCS dose and duration of OCS use prior to study were covariates; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.702 to 2.157]

2. Secondary Outcome: Percentage of Participants Achieving a >=50% Reduction in OCS Dose at Weeks 20-24 Compared to Baseline While Maintaining Asthma Control
Description: Percentage of patients whose OCS dose at weeks 20-24 was reduced >=50% compared to baseline while maintaining asthma control.
  Patients listed as "no" did not achieve the 50% reduction in baseline OCS dose goal, or did achieve that goal but lost asthma control during weeks 20 to 24, or discontinued from study drug.
Time Frame: Baseline (Day 1), Weeks 20-24
Population: ITT Analysis set; missing data are included as non-responders (No).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 89 | 88
percentage of participants
  Yes | 36 | 44
  No | 64 | 56
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 110 mg; As the analysis of the primary efficacy endpoint did not meet criteria for statistical significance (p≤0.05), the secondary efficacy endpoints were not interpreted inferentially according to the pre-defined hierarchy. P-values are nominal, meaning they were obtained from the analysis without adjustments to protect family-wise errors and should be interpreted with caution. Nominal p-values do not indicate treatment differences; Test type: Superiority; p = 0.234, Regression, Logistic — significance at 0.05; logistic regression model adjusted for treatment, stratification factors (age group and OCS dose group), duration of OCS use, and baseline value; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.786 to 2.683]

3. Secondary Outcome: Percentage of Participants Achieving an OCS Dose of <=5 mg at Weeks 20-24 While Maintaining Asthma Control
Description: Percentage of participants whose OCS dose at weeks 20-24 was <=5 mg and they maintained asthma control.
  Patients listed as "no" had a week 20-24 OCS dose > 5 mg, or whose OCS dose was <=5 mg at weeks 20-24 but did not maintain asthma control, or they discontinued from study drug.
Time Frame: Weeks 20-24
Population: ITT Analysis set; missing data are included as non-responders (No).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 89 | 88
percentage of participants
  Yes | 38 | 42
  No | 62 | 58
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 110 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.596, Regression, Logistic — significance at 0.05; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.631 to 2.229]

4. Secondary Outcome: Percent Change From Baseline in Daily Oral Corticosteroid (OCS) Dose During Weeks 20-24 Using a Mixed Model for Repeated Measures
Description: The baseline OCS dose is the prescribed optimized OCS dose following the OCS optimization period. Endpoint data are presented using an on-treatment approach. In this context, 'endpoint' was defined as the last observation obtained at a scheduled or qualified early termination visit during the treatment period. Weeks 20-24 data is included between the Week 20 dose and Week 24 for completed patients; last dose of study drug to 4 weeks after the last dose of study drug for patients who discontinued treatment early. Measurements collected outside of these defined timeframes are excluded from the analyses.
  The mixed model repeated measures (MMRM) included fixed effects for treatment, visit, treatment by visit interaction, age group, and OCS dose group, duration of OCS use and baseline value as covariates, and patient as a random effect. Unstructured covariance was assumed for the repeated measures.
Time Frame: Baseline (Day 1), Weeks 20-24
Population: ITT analysis population with available data using the on-treatment approach.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 83 | 84
percent change | -40.34 (17.318) | -58.08 (17.633)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 110 mg; Mixed model repeated measures (MMRM) with fixed effects for treatment, visit, treatment by visit interaction, age group, and OCS dose group, duration of OCS use and baseline value as covariates, and patient as a random effect. Unstructured covariance was assumed for the repeated measures; Test type: Superiority; p = 0.101, mixed model repeated measures (MMRM); Mean Difference (Final Values) = -17.75, 95% CI 2-sided [-38.986 to 3.494], Standard Error of Mean 10.759 — Reslizumab - Placebo

5. Secondary Outcome: Percentage of Participants Achieving a >=5 mg Reduction in OCS Dose at Weeks 20-24 Compared to Baseline While Maintaining Asthma Control
Description: Percentage of participants whose OCS dose at weeks 20-24 was reduced by at least 5mg from baseline and maintained asthma control. Patients listed as "no" had a week 20-24 OCS dose that did not meet the threshold of a 5mg reduction, or whose OCS dose met the threshold but did not maintain asthma control, or discontinued from study drug.
Time Frame: Baseline (Day 1), Weeks 20-24
Population: ITT Analysis set; missing data are included as non-responders (No).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 89 | 88
percentage of participants
  Yes | 35 | 41
  No | 65 | 59
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 110 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.341, Regression, Logistic — significance at 0.05; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.722 to 2.562]

6. Secondary Outcome: Annualized Rate of Clinical Asthma Exacerbations (CAEs)
Description: The annual exacerbation rate is based on clinical asthma exacerbations reported by the investigator in the eCRF.
Time Frame: Day 1 through Week 24
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: CAEs / year
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 89 | 88
CAEs / year | 1.86 [1.283 to 2.682] | 1.51 [1.052 to 2.177]
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 110 mg; Test type: Superiority; p = 0.407, Negative binomial regression model; Negative binomial regression model adjusted for stratification factors (OCS dose group), age, number of prior exacerbations, and an offset variable; CAE rate ratio = 0.82, 95% CI 2-sided [0.504 to 1.321] — reslizumab vs placebo

7. Secondary Outcome: Percentage of Participants Achieving an OCS Dose of 0 mg at Weeks 20-24 While Maintaining Asthma Control
Description: Percentage of participants who discontinue use of OCS during weeks 20-24 while maintaining asthma control.
  Patients listed as "no" continued to use OCS during weeks 20-24, or who discontinued use of OCS during weeks 20-24 but lost control of their asthma, or discontinued from study drug.
Time Frame: Weeks 20-24
Population: ITT Analysis set; missing data are included as non-responders (No).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 89 | 88
percentage of participants
  Yes | 22 | 20
  No | 78 | 80
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 110 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.628, Regression, Logistic — significance at 0.05; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.371 to 1.818]

8. Secondary Outcome: Participants With Treatment-Emergent Anti-Drug Antibody (ADA) Responses
Description: Treatment-emergent responses were defined as a positive sample post-baseline (negative baseline) OR a titer increase of >=4-fold relative to a positive baseline sample.
  Two types of antibody assay were performed, an immunogenicity status assay (ADA) and neutralizing assay (NAb).
  The ADA assay produces a positive or negative result. For samples with a positive result, a neutralizing assay was performed, which also produces a positive or negative result.
Time Frame: Weeks 4, 8, 12, 24 or early withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 89 | 88
Participants
  Positive ADA samples | 0 | 11
  Positive Nab samples | 0 | 0

9. Secondary Outcome: Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a patient administered a pharmaceutical product, regardless of whether it has a causal relationship with this treatment. In this study, asthma exacerbations (which are efficacy parameters) should not be recorded as adverse events unless assessed by the investigator as more severe than the patient's usual disease course. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
  Treatment-related adverse events or adverse events related to OCS use included events with missing relationship to study drug or OCS use, respectively.
Time Frame: Day 1 up to Week 24 (end of treatment visit); Data were included between Day 1 and Week 24 for completed patients, and Day 1 and 4 weeks after the last dose of study drug for patients who discontinued treatment early.
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 89 | 88
Participants
  Any AE | 47 | 57
  Treatment-related AE | 3 | 7
  Serious AE (SAE) | 4 | 10
  Treatment-related SAE | 0 | 0
  SAE resulting in death | 0 | 1
  AE leading to treatment discontinuation | 1 | 0
  AE related to OCS withdrawal | 2 | 3
  AE related to OCS use | 2 | 5

ADVERSE EVENTS:
Time Frame: Day 1 to Week 24
Arm/Group | Placebo | Reslizumab 110 mg
All-Cause Mortality (participants affected / at risk) | 0/89 | 1/88
Serious Adverse Events (participants affected / at risk) | 4/89 | 10/88
Other Adverse Events (participants affected / at risk) | 20/89 | 20/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=89) | Reslizumab 110 mg (N=88)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=89) | Reslizumab 110 mg (N=88)
Bronchitis (Infections and infestations) | 4 (4) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5) | 11 (13)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 5 (6)
Hypertension (Vascular disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT02501629/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT02501629/SAP_001.pdf